CLINICAL TRIAL: NCT01901978
Title: Study to Investigate Benefits of Weight Loss in Yound Adults and Adolescents
Brief Title: Study to Investigate Benefits of Weight Loss in Young Adults and Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 1007007067; R01HD040787 (NIH)
Record Dates: First submitted 2013-07-15; First posted 2013-07-17 (Estimated); Last update posted 2020-03-02 (Actual); Status verified 2020-02

CONDITIONS: Obesity; Insulin Resistance
Keywords: Obesity; Insulin Resistance; Weight loss; Women
MeSH Terms: conditions — Obesity; Insulin Resistance; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Weight Loss (Experimental): Caloric restrictive diet
  Interventions: Behavioral: Caloric restrictive diet

INTERVENTIONS:
Behavioral: Caloric restrictive diet — Patients will meet weekly with a registered dietician.

SUMMARY:
The purpose of this study is to investigate the changes in subcutaneous adipocyte size, number and gene expression after weight loss and to assess whether those changes contribute to decreases in ectopic fat accumulation and insulin resistance in women between ages of 16-32.

DETAILED DESCRIPTION:
There are no studies in young women that have prospectively studied changes in fat cell size, gene expression and insulin sensitivity during the transition from overweight/obese to normal weight. Our preliminary data suggest that the presence of ectopic fat accumulation and insulin resistance in obese children could be considered an "early phase" in the development of T2DM. We hypothesize that a 10% weight loss will restore/improve insulin sensitivity. Furthermore, we speculate that the decrease in subcutaneous fat mass after weight loss is due to a decrease in mean adipocyte cell size, but not cell number.

ELIGIBILITY:
Inclusion Criteria:

* Women ages 16-32

Exclusion Criteria:

* They will not be on any medications that are known to alter glucose or insulin metabolism, such as oral steroids, or certain psychiatric medications, such as Xeleca, Lithium and Paxil. Patients on diuretics will be excluded.

Ages: 16 Years to 32 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 14 (Actual)
Dates: Start 2011-05 (Actual); Primary Completion 2014-07 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Abdominal fat re-distribution with weight loss | 12 weeks
  To assess in young women, the effects of weight loss on abdominal fat distribution.

SECONDARY OUTCOMES:
Adipocyte cell size distrubtion and gene expression | 12 week
  With 10% weight loss, assess changes in cell size distribution and gene expression of adipocytes from the subcutaneous adipose depot.

CONTACTS AND LOCATIONS:
Overall Officials: Sonia Caprio, MD, Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD will not be shared with other researchers. Only group data that is used in data analysis for manuscripts will be shared and that is de-identified.